CLINICAL TRIAL: NCT01167283
Title: Effect of Electromyostimulation in Severe Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Electrostimulation in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: ExaEMS2005
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre Hospitalier Régional Universitaire Montpellier (Other)
Responsible Party: Prefaut/PU-PH, AEROBIE
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: APARD
Record Dates: First submitted 2010-07-13; First posted 2010-07-22 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrostimulation (Active Comparator): Neuromuscular electrical stimulation
  Interventions: Device: Electrostimulation
- Sham stimulation (Sham Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Electrostimulation — Electrostimulation: 35 Hz, 0.4 ms, 1 h; 5 times/week
  Other Names: NMES
  Arms: Electrostimulation
Device: Sham stimulation — Sham stimulation: 1 h; 5 times/week
  Other Names: Sham
  Arms: Sham stimulation

SUMMARY:
This study was designed to test the following hypothesis:

To investigate whether COPD muscles can respond to stimuli in terms of changes in fiber-type distribution.

DETAILED DESCRIPTION:
Background: Muscle dysfunction is a major problem in chronic obstructive pulmonary disease (COPD). It is characterized by muscle fiber-type redistribution and oxidative stress. Classical training does not improve these features.

Objectives: To investigate whether electrostimulation program following exacerbation can modify muscle structure and function in COPD patients.

Method: We propose to conduct a controlled and randomized clinical trial comparing the efficacy of muscle electrostimulation training of the lower limbs to sham training in 15 patients with COPD. Patients are included in either 6 weeks of electrostimulation training (active treatment group) or 6 weeks of sham electrostimulation. Primary outcomes were changes in muscle structure, muscle oxidative stress and their relationship with quadriceps force and exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients during or after exacerbation

Exclusion Criteria:

* Comorbidities that could limit exercise training
* Obesity (body mass index [BMI] > 30 kg/m²)
* Neuromuscular disease
* Pacemaker implantation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Fiber-type distribution | 6 to 8 weeks
  Typology was evaluated by immunohistochemistry

SECONDARY OUTCOMES:
Change in the strength of the quadriceps over the 6-week electrostimulation program | 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olivier OJ Jonquet, PU-PH, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France